CLINICAL TRIAL: NCT03830346
Title: Instrument-assisted Soft Tissue Mobilization and Stretching in CrossFitters
Brief Title: Instrument-assisted Soft Tissue Mobilization in CrossFitters
Acronym: MJ-IASTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MJ-IASTM
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Sports Physical Therapy
Keywords: Instrument Assisted Soft Tissue Mobilization; Manual Therapy; Muscle Stretching Exercises; Range of motion; Shoulder Joint; CrossFit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): In the experimental group, instrument-assisted soft tissue mobilization techniques and post-isometric horizontal adduction stretches were performed. The technique lasted 20 seconds in a parallel direction and 20 seconds in a perpendicular direction on the posterior shoulder and scapula muscles. While the dominant hand was used to hold the instrument, the other hand was used to tighten the skin medially to ensure an even area of treatment.
  Interventions: Other: Instrument-assisted
- Control (Experimental): Control group only underwent soft tissue mobilization. With the subject in the supine position, passively adducting the arm horizontally until the first motion barrier and performing active horizontal abduction for 5 seconds at 25% of force. The arm was then taken to the new motion barrier, repeating this process three times.
  Interventions: Other: Instrument-assisted

INTERVENTIONS:
Other: Instrument-assisted — instrument-assisted soft tissue mobilization techniques (applied with the subject in prone position. The technique lasted 20 seconds in a parallel direction and 20 seconds in a perpendicular direction on the posterior shoulder and scapula muscles. While the dominant hand was used to hold the instrument, the other hand was used to tighten the skin medially to ensure an even area of treatment) and post-isometric horizontal adduction stretches (carried out with the subject in the supine position, passively adducting the arm horizontally until the first motion barrier and performing active horizontal abduction for 5 seconds at 25% of force. The arm was then taken to the new motion barrier, repeating this process three times).

SUMMARY:
Objective. To determine the effectiveness of instrument assisted soft tissue mobilization and horizontal adduction stretch in CrossFit practitioners' shoulders.

Setting: Acero CrossFit center, city of Toledo (Spain) Design: Randomized, single-blind pilot study, with follow-up period. Participants: Twenty-one subjects of both sexes, being regular CrossFitters and in the age range of 18 to 40 years.

Intervention: The experimental group (n = 11) received 30 seconds of stretching with isometric contraction of 5 seconds and instrument assisted soft tissue mobilization. The control group (n = 10) received only 40 seconds of instrument assisted soft tissue mobilization. Each session lasted 2 to 5 minutes, 2 days a week, over a period of 4 weeks, prior to each workout.

Main Outcome measures: Shoulder internal rotation and horizontal adduction (digital inclinometer), and posterior shoulder stretch perception (Park scale) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes
* Being regular CrossFitters (workouts at least two days a week)
* In the age range of 18 to 40 years

Exclusion Criteria:

* Had suffered a shoulder injury in the 3 months prior to the study
* Had undergone shoulder surgery in the previous six months
* Had a non-attendance rate of over 15% of the intervention sessions (2 sessions)
* Had not signed the informed consent document

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline internal rotation and horizontal adduction of the shoulder after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The patient was placed in the supine position at 90º shoulder abduction, 90º elbow flexion. By stabilizing the scapula at the acromion, the shoulder was taken at a maximum range of internal rotation. The range of motion was measured with a digital inclinometer, model Tacklife MDP01, the angle of the edge of the ulna coinciding with a line perpendicular to the stretcher. For horizontal adduction, the arm was placed in the same initial position in neutral rotation and while stabilizing the lateral edge of the scapula, the arm was adducted to its maximum range of motion. The angle between the line of the ventral edge of the humerus and a line perpendicular to the stretcher was measured with the inclinometer. The range of movement in internal rotation is 0-70º and the range in horizontal adduction is 0-30º (higher degrees, greater mobility in horizontal adduction of the shoulder).

SECONDARY OUTCOMES:
Change from baseline perception of stretch after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  An 11-point numerical rating scale was used to rate subjects' perceptions of discomfort at the posterior aspect of the shoulder. This 11-point scale evaluates the discomfort from least to most, asking each subject to define the level of discomfort in the back of the shoulder in the maximum range of motion of internal rotation and horizontal adduction of the shoulder. This 11-point scale measures the perception of stretching, in a range of 0 to 10 points ("0" on the stretch sensation scale indicated ''no discomfort'' and "10" indicated ''the worst possible discomfort and increased sensitivity')

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Real Fundación Victoria Eugenia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No